CLINICAL TRIAL: NCT04473391
Title: Instrumental Gait Analysis on People With Stroke After Rehabilitation With a Synchronized FES and Cycle Ergometer System
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Corporación de Rehabilitación Club de Leones Cruz del Sur (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CorporacionRCLCS0004
Record Dates: First submitted 2020-07-13; First posted 2020-07-16 (Actual); Last update posted 2020-07-16 (Actual); Status verified 2020-07

CONDITIONS: Stroke
Keywords: Stroke; Hemiparesis; Gait; Functional Electrical Stimulation; Rehabilitation; Gait Deviation Index
MeSH Terms: conditions — Stroke; Paresis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Robot-assisted Rehabilitation (Experimental): Participants will receive Functional Electrical Stimulation (FES) training with a lower extremity cycle-ergometer (MOTOmed Viva 2, Reck GmbH., Germany) and a 6-channel FES Device (TrainFES, Biomedical Devices SpA, Chile). Patients will perform lower limb exercises assisted by the device. Training involve 24 sessions, 3 sessions per week for 8 weeks, each lasting about 45 minutes.
  Interventions: Device: Cycle-ergometer training assisted by FES for lower extremities

INTERVENTIONS:
Device: Cycle-ergometer training assisted by FES for lower extremities — The intervention consists of FES treatment sessions on a cycle ergometer for the lower extremities. Each subject received 24 sessions lasting 45 minutes each and a frequency of 3 sessions per week. The sessions will be applied by a physiotherapist with experience in electrotherapy. A 6-channel FES device (TrainFES, Biomedical Devices SpA, Chile) will be used, which consists of a stimulator unit of 95x50x30mm and 100g of weight coupled to the motorized cycle ergometer (MOTOmed Viva 2, Reck GmbH., Germany), a remote user interface consisting of an android application for the configuration of the stimulation via Bluetooth 3.1, and an inertial measurement unit positioned on the rotation axis of the cycle ergometer to detect the rotations and trigger the synchronized electrical stimulation according to the stimulation pattern pre-configured for the pedaling exercise

SUMMARY:
Functional electrical stimulation is a modality of motor rehabilitation that consists of the programmed application of bursts of electrical current to the affected neuromuscular region that aims to improve muscle strength, increase the range of motion, facilitate movement control and decrease spasticity. The present study aimed to measure the changes in the biomechanics of the gait of people with Stroke after training with functional electrical stimulation for the lower extremities.

DETAILED DESCRIPTION:
Stroke is one of the leading causes of mortality, morbidity and disability in adults in developed countries. Survivors may suffer several neurological deficits or deficiencies, such as hemiparesis, communication disorders, cognitive deficits and visuospatial perception disorders. Hemiplegia is a par loss of hemi-body voluntary motricity following a brain injury, usually resulting in alterations of the locomotor system with persistent disorders of movement and posture. Hemiplegia significantly affects gait performance. Gait recovery is an important objective in the rehabilitation program for stroke patients.The currently available treatment techniques include classical techniques of gait rehabilitation, functional electrical stimulation, electromechanic devices, robotic devices and brain-computer interfaces, among others.The evidence suggest that the combination of different rehabilitation strategies is more effective than conventional rehabilitation techniques alone. Technology-based rehabilitation methods such as robotic devices need more research to demonstrate their effects on gait recovery.

The present study aimed to identify the changes in the gait characteristics of subjects with stroke after a treatment program with FES for the lower extremities through instrumental gait analysis.

ELIGIBILITY:
Inclusion Criteria:

* unilateral lower extremity paresis
* haemorrhagic or ischemic stroke
* a minimum of six months after the acute infarction/onset of the disease
* full passive range of motion in lower extremity or at least at neutral position
* be able to stand freely
* be able to walk with or without aid for at least 20 meters in less than 2 minutes

Exclusion Criteria:

* peripheral nervous system pathology
* epilepsy
* weight over 100 kg
* no cognitive ability to follow the study instructions
* pregnancy
* use of implanted devices
* instable lower extremity joints or fixed contracture

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-03-31 (Estimated)

PRIMARY OUTCOMES:
Gait Deviation Index Baseline | Baseline
  Gait Deviation Index will be calculated for each patient using a 3D VICON infra-red camera system.
Gait Deviation Index Post-Intervention | 12 weeks
  Gait Deviation Index will be calculated for each patient using a 3D VICON infra-red camera system.

SECONDARY OUTCOMES:
Gait Speed Baseline | Baseline
  Gait Speed will be calculated for each patient using a 3D VICON infra-red camera system.
Gait Speed Post-intervention | 12 weeks
  Gait Speed will be calculated for each patient using a 3D VICON infra-red camera system.

CONTACTS AND LOCATIONS:
Overall Officials: Asterio H Andrade Gallardo, MSc., Study Chair — Corporación de Rehabilitacion Club de Leones Cruz del Sur
Locations (1):
- Corporación de Rehabilitación Club de Leones Cruz del Sur, Punta Arenas, Region of Magallanes, Chile

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Flansbjer UB, Holmback AM, Downham D, Patten C, Lexell J. Reliability of gait performance tests in men and women with hemiparesis after stroke. J Rehabil Med. 2005 Mar;37(2):75-82. doi: 10.1080/16501970410017215. PMID 15788341
- [Background] Belda-Lois JM, Mena-del Horno S, Bermejo-Bosch I, Moreno JC, Pons JL, Farina D, Iosa M, Molinari M, Tamburella F, Ramos A, Caria A, Solis-Escalante T, Brunner C, Rea M. Rehabilitation of gait after stroke: a review towards a top-down approach. J Neuroeng Rehabil. 2011 Dec 13;8:66. doi: 10.1186/1743-0003-8-66. PMID 22165907
- [Background] Gage JR. Gait analysis. An essential tool in the treatment of cerebral palsy. Clin Orthop Relat Res. 1993 Mar;(288):126-34. PMID 8458125
- [Background] Schwartz MH, Rozumalski A. The Gait Deviation Index: a new comprehensive index of gait pathology. Gait Posture. 2008 Oct;28(3):351-7. doi: 10.1016/j.gaitpost.2008.05.001. Epub 2008 Jun 18. PMID 18565753
- [Background] Popovic DB, Sinkaer T, Popovic MB. Electrical stimulation as a means for achieving recovery of function in stroke patients. NeuroRehabilitation. 2009;25(1):45-58. doi: 10.3233/NRE-2009-0498. PMID 19713618